CLINICAL TRIAL: NCT02628678
Title: An Open-label Study to Evaluate the Effect of Diet on the Tolerability of FOS, a Commercially Available Prebiotic, in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Diet on the Tolerability of FOS in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: G006-HU-PD
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Prebiotic; FOS; fructooligosaccharide; polyglycan; microbiome; microbiota; Healthy Volunteers

ARMS (1):
- Fructooligosaccharide (FOS) (Other): Subjects will be required to take 8 grams of FOS per day for a total of 10 days.
  Interventions: Dietary Supplement: FOS

INTERVENTIONS:
Dietary Supplement: FOS

SUMMARY:
The primary objective of this study is to determine the 5-day tolerability of one commercially available prebiotic food ingredient, FOS, in healthy human subjects with and without diet control.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent;
2. Be male or female of any race, between 18 and 65 years of age;
3. Have a BMI > 20 & < 27 kg/m2;
4. Be willing to follow a controlled low fiber diet for a period of 11 days;

Exclusion Criteria:

1. Are less than 18 and greater than 65 years of age;
2. Are hypersensitive to any of the components of FOS;
3. Are currently taking probiotic or prebiotic supplements, or have taken them in the past 28 days;
4. Unwilling to avoid probiotics/prebiotics supplements for the duration of the study;
5. Have a significant acute or chronic, unstable and untreated disease or any condition which contraindicates, in the investigators judgment, entry to the study;
6. Subject is a smoker;
7. Subject has a history of drug and/or alcohol abuse at the time of enrollment;
8. Taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results;
9. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
10. Subjects may not be receiving treatment involving experimental drugs;
11. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | 22 days

SECONDARY OUTCOMES:
The effect of controlling diet on the tolerability of FOS by analyzing the gut microbiome | 22 days

OTHER OUTCOMES:
The effect of FOS on each subject's gut microbiome | 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- Kaleido Biosciences, Cambridge, Massachusetts, United States